CLINICAL TRIAL: NCT00670878
Title: Prospectively Randomized Phase III Trial, Studying the Benefits of Adjuvant Sequential vs. Combined Taxane Based Chemotherapy, Followed by Different Biological Treatment Strategies in Early, HER2-positive Breast Cancer
Brief Title: Studying the Benefits of Adjuvant Sequential vs. Combined Taxane Based Chemotherapy, Followed by Different Biological Treatment Strategies in Early, HER2-positive Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Philip Hepp, study doctor, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SUCCESS-B
Record Dates: First submitted 2008-04-30; First posted 2008-05-02 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-03

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: 3 x FEC 3 x DOC / Gemcitabine
- B (Active Comparator)
  Interventions: Drug: 3 x FEC 3 x DOC

INTERVENTIONS:
Drug: 3 x FEC 3 x DOC / Gemcitabine — 3 cycles of 5-Fluorouracil 500 mg/m² i.v. body surface area and Epirubicin 100 mg/m² i.v. and Cyclophosphamide 500 mg/m² i.v., (FEC100), each administered on day 1, repeated on day 22, subsequently followed by 3 cycles of Docetaxel 75 mg/m² body surface area i.v. (D), and Gemcitabine 1000 mg/m² i.v. (30 min infusion) (G), administered on day 1, followed by Gemcitabine 1000 mg/m² i.v. (30 min infusion) on day 8, repeated on day 22
  Arms: A
Drug: 3 x FEC 3 x DOC — 3 cycles of 5-Fluorouracil 500 mg/m² i.v. body surface area and Epirubicin 100 mg/m² i.v. and Cyclophosphamide 500 mg/m² i.v., (FEC100), each administered on day 1, repeated on day 22, subsequently followed by 3 cycles of Docetaxel 100 mg/m² body surface area i.v. (D), administered on day 1, repeated on day 22
  Arms: B

SUMMARY:
This is an open-label, multicenter randomized controlled, Phase III study comparing the disease free survival after randomisation in patients treated with 3 cycles of Epirubicin-Fluorouracil-Cyclophosphamide (FEC)-chemotherapy, followed by 3 cycles of Docetaxel (D)-chemotherapy versus 3 cycles of Epirubicin-Fluorouracil- Cyclophosphamide (FEC), followed by 3 cycles of Gemcitabine-Docetaxel(DG)- chemotherapy. Patients will be required to have HER2-neu positive disease and histopathological proof of axillary lymph node metastases (pN1-3) or high risk node negative, defined as: pT>=2 or histopathological grade 3, or age <= 35 or negative hormone receptor', but are not allowed to have evidence of distant disease. Patients will have to be entered into the study no later than 6 weeks after complete resection of the primary tumor. No other antineoplastic treatment other than surgical treatment, the defined cytotoxic and endocrine treatment and radiotherapy will be allowed prior to study entry and during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

* Primary epithelial invasive carcinoma of the breast pT1-4, pN0-3, M0
* Evidence of HER2-neu overexpressing (IHC +++) or amplifying (FISH +) tumor
* Histopathological proof of axillary lymph node metastases (pN1-3) or high risk node negative, defined as at least two criteria of the following: 'pT³2, histopathological grade 3, age £ 35, negative hormone receptor'
* Complete resection of the primary tumor with margins of resection free of invasive carcinoma not more than 6 weeks ago
* Females >= 18 years of age
* Performance Status <2 on ECOG-Scale
* Adequate bone marrow reserve: leucocytes ³ 3.0 x 109/l and platelets ³ 100 x 109/l
* Bilirubin within one fold of the reference laboratory's normal range, ASAT (SGOT), ALAT (SGPT) and AP within 1,5 fold of the reference laboratory's normal range for patients
* Intention of regular follow up visits for the duration of the study
* Ability to understand the nature of the study and to give written informed consent
* Women of childbearing potential must agree to use an effective method of contraception (Pearl-Index < 1, e.g. , intrauterine devices or sterilization) during treatment and for at least 6 months thereafter.

Exclusion Criteria:

* Inflammatory breast cancer
* Previous or concomitant cytotoxic or other systemic antineoplastic treatment which is not part of this study
* A second primary malignancy (except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin)
* Cardiomyopathy with impaired ventricular function (NYHA > II), cardiac arrhythmias influencing LVEF and requiring medication, history of myocardial infarction or angina pectoris within the last 6 months, or arterial hypertension not being controlled by medication
* Any known hypersensitivity reaction against docetaxel, epirubicin, cyclophosphamide, gemcitabine or any other medication included in the study protocol. The contraindication, warning notices and measures of precaution of the products, as notified in the product information, have to be respected
* Instable diabetes mellitus, out of sufficient medical control
* Use of any investigational agent within 3 weeks prior to inclusion
* Patients in pregnancy or breast feeding (in premenopausal women contraception has to be assured)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 799 (Estimated)
Dates: Start 2008-06; Primary Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Disease free survival | 5 y

SECONDARY OUTCOMES:
Overall survival time after randomization | 5 Y
Distant disease free survival | 5 Y
Toxicity | 5 Y
Changes in quality of life over time as defined by EORTC QLQ-C30 and QLQBR23 questionnaire | 5 Y
Skeletal related events | 5 Y
Incidence of secondary primaries | 5 Y
Endpoints of adjunct translational research program | 5 Y

CONTACTS AND LOCATIONS:
Locations (1):
- Frauenklinik der Universität München Campus Innenstadt, Munich, Germany

REFERENCES:
- See also: Related Info — http://www.success-studie.de